CLINICAL TRIAL: NCT01527487
Title: A Randomized Phase II Study of Eribulin/Cyclophosphamide or Docetaxel/Cyclophosphamide as Neoadjuvant Therapy in Locally Advanced HER2-Negative Breast Cancer
Brief Title: Trial of Eribulin/Cyclophosphamide or Docetaxel/Cyclophosphamide as Neoadjuvant Therapy in Locally Advanced HER2-Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 197
Record Dates: First submitted 2012-01-31; First posted 2012-02-07 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-10

CONDITIONS: HER2 Negative Breast Cancer
Keywords: breast cancer; eribulin; Halaven; taxotere
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eribulin+Cyclophosphamide (ErC) (Experimental): Eribulin (Er): 1.4mg/m2 IV (Days 1 and 8) given short (≤1.5 minutes) IV infusion, per institutional standard
  Cyclophosphamide (C): 600 mg/m2 IV (Day 1), given by IV infusion, per institutional standard
  Interventions: Drug: Eribulin; Drug: Cyclophosphamide
- Docetaxel+Cyclophosphamide (TC) (Experimental): Docetaxel (T): 75 mg/m2 IV (Day 1), given by 1-hour IV infusion
  Cyclophosphamide (C): 600 mg/m2 IV (Day 1), given by IV infusion, per institutional standard
  Interventions: Drug: Cyclophosphamide; Drug: Docetaxel

INTERVENTIONS:
Drug: Eribulin — 1.4 mg/m2 IV (Days 1 & 8), given short (≤15 minute) IV infusion, per institutional standard
  Other Names: Halaven
  Arms: Eribulin+Cyclophosphamide (ErC)
Drug: Cyclophosphamide — Cyclophosphamide will be given as an IV infusion (600 mg/m2) on Day 1 of each treatment cycle over approximately 30 minutes, or per institutional standard.
  Other Names: Cytoxan
Drug: Docetaxel — Patients assigned to Treatment Arm 2 will receive docetaxel 75 mg/m2 IV on Day 1 of each treatment cycle every 3 weeks.
  Other Names: Taxotere
  Arms: Docetaxel+Cyclophosphamide (TC)

SUMMARY:
The investigators propose a randomized phase II study evaluating the pCR and toxicity profiles of combination eribulin/cyclophosphamide (ErC) and docetaxel /cyclophosphamide (TC) as neoadjuvant therapy for locally advanced HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive adenocarcinoma of the breast.
2. Primary palpable disease confined to the breast and axilla on physical examination (clinical Stage II or III disease). For patients without clinically suspicious axillary adenopathy, the primary must be >2 cm in diameter by physical examination or imaging studies (clinical T2-3, N0-2, M0). For patients with clinically suspicious axillary adenopathy, the primary breast tumor can be any size (clinical T1-3, N1-2, M0). Patients who have had axillary node dissection and have pN3a (i.e. ≥10 involved axillary nodes) are also eligible.
3. Patients entering the trial after undergoing an axillary node dissection will be eligible if they meet other entry criteria.
4. Estrogen receptor (ER) and progesterone receptor (PR) status in the primary tumor known or pending at the time of study registration.
5. Resolution of all acute effects of surgical procedures to ≤ grade 1. For patients who had or will have, a sentinel node and/or axillary node dissection, completion at least 1 week prior to the initiation of study treatment with a well-healed wound is required.
6. Bilateral, synchronous breast cancer is allowed if both primary tumors are HER2-negative and at least one meets the specified qualifying tumor or nodal inclusion criteria.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-2.
8. Patients entering this study must be willing to provide release of tumor tissue collected at baseline during a diagnostic procedure if available, and at the time of future surgical procedure(s) for correlative testing. If tissue is not available, the patient will still be eligible for enrollment to the study.
9. No evidence of metastatic disease, as documented by complete staging workup ≤8 weeks prior to initiation of study treatment.
10. No prior treatment for this breast cancer with the exception of criterion #3.
11. HER2-negative tumor status defined as:

    * Immunohistochemical (IHC) 0-1+ or
    * IHC 2+ or IHC 3+ confirmed as FISH (Fluorescence in situ hybridization) or SISH (Silver in situ hybridization) negative (defined by ratio <2.2)
12. Adequate hematologic function defined as:

    * Absolute neutrophil count (ANC) ≥1500/μL
    * Hemoglobin (Hgb) ≥10 g/dL
    * Platelets ≥100,000/uL
13. Adequate liver function defined as:

    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x the upper limit of normal (ULN)
    * Total bilirubin ≤ the institutional ULN
14. Adequate renal function defined as:

    * Serum creatinine ≤1.5 mg/dL x ULN OR calculated creatinine clearance ≥50 mL/min by the Cockcroft-Gault method:

    GRF =(140-age) x (weight/kg) x (0.85 if female) (72 x serum creatinine mg/dL)
15. Other laboratory testing:

    * Serum magnesium ≥ the institutional lower limit of normal (LLN)
    * Serum potassium ≥the institutional LLN
16. Female and ≥18 years of age.
17. Negative serum pregnancy test within <7 days prior to initial trial treatment.
18. Female patients who are not of child-bearing potential, and female patients of child-bearing potential who agree to use adequate contraceptive measures that are approved by their study physician while receiving study treatment and continuing for 3 weeks after the last dose of study drug treatment, who are not breastfeeding, and who have a negative serum pregnancy test prior to start of dosing.
19. Willingness and ability to comply with trial and follow-up procedures.
20. Ability to understand the nature of this trial and give written informed consent.

Exclusion Criteria:

1. Clinical T4 lesions, including inflammatory breast cancer. Clinical N3 involvement (e.g., ipsilateral, infraclavicular, supraclavicular, and internal mammary nodes).
2. Peripheral neuropathy (motor or sensory) > grade 1 according to Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0).
3. Patient has received radiotherapy for treatment of previous cancer that included ≥30% of major bone marrow containing areas (e.g., pelvis, lumbar, spine).
4. Known or suspected allergy or hypersensitivity to any of the study drugs (i.e., eribulin, cyclophosphamide, docetaxel) or known hypersensitivity to polysorbate 80.
5. Patients with acute or chronic liver or renal disease or pancreatitis.
6. Known diagnosis of human immunodeficiency virus (HIV), Hepatitis B (HBV) or Hepatitis C (HCV).
7. Concurrent treatment with an ovarian hormonal replacement therapy or with hormonal agents such as raloxifene, tamoxifen or other selective estrogen receptor modulator (SERM). Patients must have discontinued use of such agents prior to beginning study treatment. However, use of GNRH agonists for the purpose of fertility preservation or suppression of heavy menses is permitted (see Section 5.4.1).
8. Patient has any of the following cardiac diseases currently or within the last 6 months:

   * Left Ventricular Ejection Fraction (LVEF) <45% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
   * Heart rate-corrected QT interval (QTc) > 480 ms on screening electrocardiogram (ECG) (using Bazett's formula)
   * Unstable angina pectoris
   * Congestive heart failure (New York Heart Association [NYHA] ≥ Grade 2
   * Acute myocardial infarction
   * Conduction abnormality not controlled with pacemaker or medication
   * Significant ventricular or supraventricular arrhythmias (Patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible).
   * Valvular disease with significant compromise in cardiac function
9. Chronic use of drugs that cause QTc prolongation. Patients must discontinue use of these drugs 7 days prior to the start of study treatment.
10. Presence of other active cancers, or history of treatment for invasive cancer ≤5 years. Patients with stage I cancer who have received definitive local treatment at least 3 years previously, and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e. non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
11. Patients may not receive any other investigational or anti-cancer treatments while participating in this trial.
12. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
13. Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-06; Primary Completion 2014-09 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A Yardley, MD, Study Chair — SCRI Development Innovations, LLC
Locations (15):
- United States (15):
  - Florida Cancer Specialists South, Fort Myers, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - Florida Cancer Specialists North, St. Petersburg, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Mercy Hospital, Portland, Maine
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Grand Rapids Oncology Program, Grand Rapids, Michigan
  - Research Medical Center, Kansas City, Missouri
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - Oncology Hematology Care, Inc, Cincinnati, Ohio
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Virginia Cancer Institute, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This neoadjuvant trial evaluated the combination of eribulin/cyclophosphamide (ErC) versus docetaxel/cyclophosphamide (TC) in women with clinical stage II-III breast cancers. Between JUN 2012 and APR 2014, 76 patients were enrolled.
Pre-assignment Details: After a 10-patient lead-in to confirm safety and feasibility of ErC, subsequent patients (66) were randomized 2 to 1 for treatment with: (1) ErC (44 patients) or (2) TC (22 patients). Both regimens were administered every 21 days for 6 cycles followed by surgery.
Groups:
- Eribulin+Cyclophosphamide: ErC: Eribulin (Er): 1.4 mg/m^2 by IV infusion (Days 1 and 8); Cyclophosphamide (C): 600 mg/m^2 by IV infusion (Day 1)
  Administered every 21 days for 6 cycles followed by surgery.
- Docetaxel+Cyclophosphamide: TC: Docetaxel (T): 75 mg/m^2 by IV infusion (Day 1); Cyclophosphamide (C): 600 mg/m^2 by IV infusion (Day 1)tandard.
  Administered every 21 days for 6 cycles followed by surgery.
Period: Overall Study
Arm/Group | Eribulin+Cyclophosphamide: ErC | Docetaxel+Cyclophosphamide: TC
Started | 54 (Includes 10 patients from safety lead-in.) | 22
Completed | 46 (Patients who completed 6 cycles plus surgery.) | 15
Not Completed | 8 | 7
Not completed — MD Discretion/Lack of Efficacy | 3 | 4
Not completed — Disease Progression | 4 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis population for ErC includes 10 lead-in and 44 randomized patients.
Groups:
- Eribulin+Cyclophosphamide (ErC): Eribulin (Er): 1.4mg/m2 IV (Days 1 and 8) given short (≤1.5 minutes) IV infusion, per institutional standard;
  Cyclophosphamide (C): 600 mg/m2 IV (Day 1), given by IV infusion, per institutional standard
- Docetaxel+Cyclophosphamide (TC): Docetaxel (T): 75 mg/m2 IV (Day 1), given by 1-hour IV infusion;
  Cyclophosphamide (C): 600 mg/m2 IV (Day 1), given by IV infusion, per institutional standard
- Total: Total of all reporting groups
Arm/Group | Eribulin+Cyclophosphamide (ErC) | Docetaxel+Cyclophosphamide (TC) | Total
Number analyzed (Participants) | 54 | 22 | 76
Age, Continuous [Median (Full Range); unit: years] | 53 [23 to 77] | 51 [38 to 73] | 52 [23 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 22 | 76
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 22 | 76

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) Rate in Patients Treated With ErC for 6 Cycles Prior to Surgery
Description: One cycle = 21 days. Pathologic CR is defined as the absence of invasive tumor in the breast and lymph node tissue removed at the time of definitive surgery as judged by the local pathologist.
Time Frame: 18 weeks
Population: Patients who completed 6 cycles and proceeded to surgery.
Measure: Number; unit: percentage of surgical patients
Groups:
- Eribulin+Cyclophosphamide (ErC): Eribulin (Er): 1.4mg/m^2 (Days 1 and 8 of each treatment cycle) by IV infusion
  Cyclophosphamide (C): 600 mg/m^2 IV (Day 1 of each treatment cycle) by IV infusion
- Docetaxel+Cyclophosphamide (TC): Docetaxel (T): 75 mg/m^2 (Day 1 of each treatment cycle), by IV infusion
  Cyclophosphamide (C): 600 mg/m^2 (Day 1 of each treatment cycle)
Arm/Group | Eribulin+Cyclophosphamide (ErC) | Docetaxel+Cyclophosphamide (TC)
Number analyzed (Participants) | 39 | 20
percentage of surgical patients | 18 | 10

2. Secondary Outcome: The Number of Adverse Events as a Measure of Safety and Tolerability.
Description: Treatment-Related Adverse Events occurring in >= 15% of treated patients
Time Frame: 43 months
Measure: Number; unit: participants
Groups:
- Eribulin+Cyclophosphamide (ErC): Eribulin (Er): 1.4mg/m^2 (Days 1 and 8 of each treatment cycle) by IV infusion.
  Cyclophosphamide (C): 600 mg/m^2 (Day 1 of each treatment cycle) by IV infusion.
- Docetaxel+Cyclophosphamide (TC): Docetaxel (T): 75 mg/m^2 (Day 1 of each treatment cycle) by IV infusion.
  Cyclophosphamide (C): 600 mg/m^2 (Day 1 of each treatment cycle) by IV infusion.
Arm/Group | Eribulin+Cyclophosphamide (ErC) | Docetaxel+Cyclophosphamide (TC)
Number analyzed (Participants) | 54 | 22
participants
  Fatigue | 32 | 14
  Alopecia | 25 | 14
  Nausea | 26 | 8
  Peripheral Sensory Neuropathy | 18 | 10
  Neutrophil Count Decreased | 21 | 6
  Constipation | 15 | 6
  Diarrhea | 11 | 10
  Anemia | 12 | 8
  Headache | 9 | 4
  Dysgeusia | 8 | 5
  White Blood Cell Decreased | 8 | 5
  Myalgia | 7 | 6
  Hot Flashes | 7 | 3
  Mucositis | 5 | 5
  Arthralgia | 2 | 8
  Edema Limbs | 2 | 8

3. Secondary Outcome: Clinical Response Rate (cRR) of ErC as Neoadjuvant Therapy
Description: Defined as the number of patients with a best response of clinical complete or partial response (cCR or cPR) divided by the number of patients qualified for tumor response analysis per Response Evaluation Criteria in Solid Tumors Criteria (RECIST) v1.1 for target lesions and assessed by MRI or CT. Complete Response (CR) defined as disappearance of all target lesions; Partial Response (PR) defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD;
Time Frame: 43 months
Population: All patients evaluated/evaluable per RECIST v1.1
Measure: Number; unit: percentage of participants
Groups:
- Eribulin+Cyclophosphamide (ErC): Eribulin (Er): 1.4mg/m^2 (Days 1 and 8 of each treatment cycle) by IV infusion.
  Cyclophosphamide (C): 600 mg/m^2 IV (Day 1 of each treatment cycle) by IV infusion.
Arm/Group | Eribulin+Cyclophosphamide (ErC) | Docetaxel+Cyclophosphamide (TC)
Number analyzed (Participants) | 34 | 17
percentage of participants | 67.6 | 64.7

4. Secondary Outcome: Disease-Free Survival (DFS) at 2 Years
Description: Defined as the percent probability that participants had not experienced disease recurrence or died from any cause at 2 years post-surgery, analyzed by Kaplan-Meier methodology.
Time Frame: 24 months
Population: Includes all patients that completed surgery.
Measure: Number (95% Confidence Interval); unit: percent probability of survival
Groups:
- Eribulin+Cyclophosphamide (ErC): Eribulin (Er): 1.4mg/m^2 IV (Days 1 and 8 of each treatment cycle) by IV infusion.
  Cyclophosphamide (C): 600 mg/m^2 IV (Day 1 of each treatment cycle by IV infusion.
- Docetaxel+Cyclophosphamide (TC): Docetaxel (T): 75 mg/m2 IV (Day 1), given by 1-hour IV infusion
  Cyclophosphamide (C): 600 mg/m2 IV (Day 1), given by IV infusion, per institutional standard
  Cyclophosphamide: Cyclophosphamide will be given as an IV infusion (600 mg/m2) on Day 1 of each treatment cycle over approximately 30 minutes, or per institutional standard.
  Docetaxel: Patients assigned to Treatment Arm 2 will receive docetaxel 75 mg/m2 IV on Day 1 of each treatment cycle every 3 weeks.
Arm/Group | Eribulin+Cyclophosphamide (ErC) | Docetaxel+Cyclophosphamide (TC)
Number analyzed (Participants) | 53 | 21
percent probability of survival | 82.35 [60.15 to 92.85] | 89.06 [62.66 to 97.17]

ADVERSE EVENTS:
Time Frame: 43 months
Groups:
- Eribulin+Cyclophosphamide (ErC): Eribulin (Er): 1.4mg/m2 IV (Days 1 and 8) given short (≤1.5 minutes) IV infusion, per institutional standard
  Cyclophosphamide (C): 600 mg/m2 IV (Day 1), given by IV infusion, per institutional standard
  Eribulin: 1.4 mg/m2 IV (Days 1 & 8), given short (≤15 minute) IV infusion, per institutional standard
  Cyclophosphamide: Cyclophosphamide will be given as an IV infusion (600 mg/m2) on Day 1 of each treatment cycle over approximately 30 minutes, or per institutional standard.
Arm/Group | Eribulin+Cyclophosphamide (ErC) | Docetaxel+Cyclophosphamide (TC)
Serious Adverse Events (participants affected / at risk) | 4/54 | 2/22
Other Adverse Events (participants affected / at risk) | 44/54 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin+Cyclophosphamide (ErC) (N=54) | Docetaxel+Cyclophosphamide (TC) (N=22)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Sepsis (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin+Cyclophosphamide (ErC) (N=54) | Docetaxel+Cyclophosphamide (TC) (N=22)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 32 | 14
ANEMIA (Blood and lymphatic system disorders) | 18 | 8
ANOREXIA (Metabolism and nutrition disorders) | 3 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 8
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 0
ASTHENIA (General disorders) | 4 | 1
CHILLS (General disorders) | 3 | 0
CONSTIPATION (Gastrointestinal disorders) | 16 | 6
DIARRHEA (Gastrointestinal disorders) | 12 | 10
DIZZINESS (Nervous system disorders) | 5 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 | 0
DYSGEUSIA (Nervous system disorders) | 7 | 4
DYSPEPSIA (Gastrointestinal disorders) | 9 | 0
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 4 | 2
EDEMA (General disorders) | 3 | 8
FATIGUE (General disorders) | 40 | 14
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 0
FEVER (General disorders) | 6 | 1
HEADACHE (Nervous system disorders) | 11 | 4
HOT FLASHES (General disorders) | 9 | 3
INSOMNIA (Nervous system disorders) | 5 | 3
LEUKOPENIA (Blood and lymphatic system disorders) | 15 | 5
LYMPHOCYTE COUNT DECREASED (Investigations) | 3 | 0
MALAISE (General disorders) | 3 | 0
MUCOSITIS (Gastrointestinal disorders) | 6 | 5
MYALGIA (Musculoskeletal and connective tissue disorders) | 9 | 6
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 2 | 2
NAIL DISCOLORATION (Skin and subcutaneous tissue disorders) | 1 | 3
NAUSEA (Gastrointestinal disorders) | 33 | 8
NEUTROPENIA (Blood and lymphatic system disorders) | 26 | 5
PARESTHESIA (Nervous system disorders) | 5 | 0
PERIPHERAL NEUROPATHY (Nervous system disorders) | 19 | 10
POST NASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 3 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 0
RASH (Skin and subcutaneous tissue disorders) | 5 | 2
SCALP PAIN (Skin and subcutaneous tissue disorders) | 0 | 2
TASTE ALTERATION (Nervous system disorders) | 5 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 | 1
URINARY TRACT INFECTION (Renal and urinary disorders) | 3 | 0
VOMITING (Gastrointestinal disorders) | 3 | 0
WATERING EYES (Eye disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites